CLINICAL TRIAL: NCT06453616
Title: Cluster Randomized Controlled Trial Evaluating the Effectiveness of the "Hello Bundle" Intervention in Reducing Burnout Among ICU Healthcare Professionals
Brief Title: Evaluating the Effectiveness of the "Hello Bundle" Intervention in Reducing Burnout Among ICU Healthcare Professionals
Acronym: HELLO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Society of Intensive Care Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HELLO
Record Dates: First submitted 2024-05-18; First posted 2024-06-11 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Prevalence of Burn-out Among Intensive Care Professionals
Keywords: Burn-out; Healthcare professionals; Job leave intent; Ethical climate; Intensive care medicine
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: cluster randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The methodologists will be blind of the study group and not aware on whether group A and B are control or intervention groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Hello arm (Intervention arm) (Experimental): The intervention arms will receive the Hello Bundle (posters, email reminders, morning huddles, hello jar, hello board and a led example).
  The bundle includes six components: displaying Hello posters all over the ICU, email reminders every week to study investigators (4 times for the 4 week study period), inciting Hello during morning huddles, lead by example by ICU heads, Hello Jar to insert messages emphasizing well being at work and posters to allow HCP write hello messages.
  Interventions: Behavioral: Hello bundle
- The usual arm (Controlled arm) (No Intervention): No intervention will be performed in the control groups which will behave as per their standard.

INTERVENTIONS:
Behavioral: Hello bundle — Hello Bundle comprises : posters, email reminders, morning huddles, hello jar, hello board and a led example.
  Participants will have to fill out a questionnaire before and after the intervention.
  The main components of the questionnaire include respondent's characteristics, visitation policies, team-family interactions, family-centeredness (VAS), and practices at the end of life. ICU-conflicts (VAS), symptoms of burnout, and a VAS to rank the ethical climate, satisfaction with work, and intent to leave the job. Symptoms of burnout will be measured using the validated version of the 22-item Maslach Burnout Inventory (MBI, Human Services version)
  Arms: The Hello arm (Intervention arm)

SUMMARY:
Burnout among healthcare professionals in intensive care units (ICUs) is a prevalent concern with significant implications for both staff well-being and patient care outcomes. This protocol outlines a cluster randomized controlled trial designed to evaluate the effectiveness of the "Hello Bundle" intervention in reducing burnout among ICU healthcare professionals. The intervention comprises of various components aimed at fostering a positive and supportive work environment, including the distribution of Hello Campaign Posters, Email Reminders, Morning Huddles, Hello Jars, and Lead by Example initiatives. A hello board updated daily will be made available in each ICU. The trial will involve 146 participating centers affiliated with the ESICM, randomly assigned to intervention and control groups. Each center will have to include at least 50 HCP. Data will be collected from healthcare professionals at baseline, during the intervention period, and at follow-up, focusing on the prevalence of burnout, satisfaction with care, professional's intent to leave the ICU, and perceptions of the ethical climate. Statistical analysis will compare outcomes between intervention and control groups, aiming to demonstrate a reduction in the prevalence of burnout from 40% to 30% with an intra-class coefficient of 0.3 and a statistical power of 90%. This trial holds the potential to provide valuable insights into effective strategies for addressing burnout in ICU settings, ultimately benefiting both staff and patients.

DETAILED DESCRIPTION:
ESICM affiliates (those registered on the ESICM mailing list) will receive a message in May 2024 with an invitation to take part in the cluster randomized trial. Two reminders will be sent until June 2024.

In each participating ICU, a dyad of investigators (physician and a nurse) will complete the ICU questionnaire (hospital size and ICU type, university affiliated, specialized ICU) and collect the willingness of each HCP to participate in the study. Participation rate will need to be >50% to be eligible for the trial. For those who are eligible, email addresses of HCPs will be required to be able to encourage them to implement the intervention. Online consent will be obtained from all participants to take part in the study and to use the data collected in the questionnaires. HCP characteristics, including age, sex, experience, and working conditions, will be collected. The dyad of investigators in each ICU will also set up a designated "Hello Board" every day with a date where staff members can write short greetings or positive messages to each other using markers or sticky notes. This can serve as a visual reminder to greet each other and foster a sense of camaraderie among team members.

The main components of the questionnaire include respondent's characteristics, visitation policies, team-family interactions, family-centeredness (VAS), and practices at the end of life. ICU-conflicts (VAS), symptoms of burnout, and a VAS to rank the ethical climate, satisfaction with work, and intent to leave the job. Symptoms of burnout will be measured using the validated version of the 22-item Maslach Burnout Inventory (MBI, Human Services version), which includes three subscales: emotional exhaustion (9 items), depersonalization (5 items), and personal accomplishment (8 items). Each item is scored from 0 (never) to 6 (every day). Respondents with high emotional exhaustion (≥27) and/or high depersonalization (≥10) scores will be considered to have symptoms of burnout.

Visual analogue scales (VAS) are used to assess the intensity of unidimensional measures. Two anchors are provided: for 0 (no symptom/lowest rating) and 10 (the most intense symptom/highest rating). VASs are convenient, easy, and rapid to administer and have been proved reliable for measuring a characteristic, subjective phenomenon, or attitude that is believed to range across a continuum of values and cannot easily be directly measured.

It is proposed to have a cluster randomized controlled trial with 146 participating centers, randomly assigned to intervention and control groups. All centers will be affiliated with ESICM, and data will be collected from HCP without involving any patient data. The primary endpoint is the prevalence of burnout measured by the Maslach Burnout Inventory (MBI) scale, between intervention and control groups with secondary endpoints including the comparison of burn-out prevalence before and after the intervention, HCP, satisfaction with work, HCP's intent to leave the ICU, and ethical climate rank and the importance of family and patient-centered care.

Statistical Analysis Quantitative variables will be described as median (interquartile range [IQR]) and will be compared between groups using the non-parametric Wilcoxon rank-sum test. Qualitative variables will be described as frequency (percentages) and will be compared between groups using Fisher's exact test.

Primary endpoint will be prevalence of burn out as defined by a high emotional exhaustion (score, ≥27) and/or high depersonalization (score, ≥10). Secondary endpoint will include individual components of the Maslach Burn Out Inventory and VAS, as well as HCP's intent to leave the ICU and ethical climate.

Primary and secondary analyses will be performed at an individual level adjusting for clustering. No imputation will be performed for missing variables.

Subgroup analyses will be conducted to explore potential moderators of intervention effectiveness.

Statistical analyses will be performed with R statistical software, version 3.4.3 (available online at http://www.r-project.org/) and packages 'lme4',and 'lmerTest'. A p value <0.05 will be considered significant.

Sample size:

Assuming an intra-class correlation of 0.3, 146 centers and 50 respondents per center, the study would allow to demonstrate a reduction in burnout prevalence from 40% to 30% with a statistical power of 90%.

How to get 200 centers, each including 50 healthcare providers? The steering committee includes 20 persons, each inviting 4 centers = 80 ESICM executive committee and council include 30 more people, each inciting 2 ICUs: 60 Note that immediately upon acceptance, centers complete the ICU characteristics form to be published anywhere to foster the group feeling.

The "Hello Bundle" intervention will be implemented in intervention group centers over a period of 30 days. The Hello board that is updated every day and regular communication will ensure adherence to the intervention components, and centers will receive support as needed to facilitate implementation. Training sessions and educational materials will be provided to ensure staff understanding and engagement with the intervention.

To allow control centers benefit from the intervention and avoid frustration, the intervention will be made possible (but optional) in the control centers 90 days after the end of the trial, and will not be followed by other measurements.

The intervention closed in the intervention groups on November 10, 2024. The collection of the post-intervention burn-out questionnaires has started and it is set to close on 20 December 2024.

ELIGIBILITY:
Inclusion Criteria:

* healthcare professionals working in intensive care.

Exclusion Criteria:

* under 18 years of age healthcare professionals
* healthcare professionals not working in intensive care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7300 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
The number of healthcare professionals with symptoms of burnout as defined by a high emotional exhaustion and/or a high depersonalization in the Maslach Burnout inventory | 1 month
  Primary endpoint will be prevalence of burn out as defined by a high emotional exhaustion (score, ≥27) and/or high depersonalization (score, ≥10).

SECONDARY OUTCOMES:
The number of healthcare professionals with high emotional exhaustion. | 1 Month after the intervention
  When specified, the outcome will be measured using Visual Analogue Scales that assess the intensity of unidimensional measures. Two anchors are provided and respondents provide an answer that ranges between zero (minimal symptoms/negative experience) to ten (maximum symptoms/positive experience).
The number of healthcare professionals with high depersonalization. | 1 Month after the intervention
  When specified, the outcome will be measured using Visual Analogue Scales that assess the intensity of unidimensional measures. Two anchors are provided and respondents provide an answer that ranges between zero (minimal symptoms/negative experience) to ten (maximum symptoms/positive experience).
The median score of the "loss of accomplishment at work" domain of the Maslach Burnout inventory. | 1 Month after the intervention
  When specified, the outcome will be measured using Visual Analogue Scales that assess the intensity of unidimensional measures. Two anchors are provided and respondents provide an answer that ranges between zero (minimal symptoms/negative experience) to ten (maximum symptoms/positive experience).
The perception of ethical climate at work | 1 Month after the intervention
  When specified, the outcome will be measured using Visual Analogue Scales that assess the intensity of unidimensional measures. Two anchors are provided and respondents provide an answer that ranges between zero (minimal symptoms/negative experience) to ten (maximum symptoms/positive experience).
The perception of satisfaction at work | 1 Month after the intervention
  When specified, the outcome will be measured using Visual Analogue Scales that assess the intensity of unidimensional measures. Two anchors are provided and respondents provide an answer that ranges between zero (minimal symptoms/negative experience) to ten (maximum symptoms/positive experience).
The perception of professional conflicts (visual analogue scale). | 1 Month after the intervention
  When specified, the outcome will be measured using Visual Analogue Scales that assess the intensity of unidimensional measures. Two anchors are provided and respondents provide an answer that ranges between zero (minimal symptoms/negative experience) to ten (maximum symptoms/positive experience).
The intention to leave the ICU | 1 Month after the intervention
  When specified, the outcome will be measured using Visual Analogue Scales that assess the intensity of unidimensional measures. Two anchors are provided and respondents provide an answer that ranges between zero (minimal symptoms/negative experience) to ten (maximum symptoms/positive experience).
The rating of patient centered care | 1 Month after the intervention
  When specified, the outcome will be measured using Visual Analogue Scales that assess the intensity of unidimensional measures. Two anchors are provided and respondents provide an answer that ranges between zero (minimal symptoms/negative experience) to ten (maximum symptoms/positive experience).
The rating of family centered care | 1 Month after the intervention
  When specified, the outcome will be measured using Visual Analogue Scales that assess the intensity of unidimensional measures. Two anchors are provided and respondents provide an answer that ranges between zero (minimal symptoms/negative experience) to ten (maximum symptoms/positive experience).
The proportion of burnout before and after the intervention (in the intervention cluster) | 1 Month after the intervention
  When specified, the outcome will be measured using Visual Analogue Scales that assess the intensity of unidimensional measures. Two anchors are provided and respondents provide an answer that ranges between zero (minimal symptoms/negative experience) to ten (maximum symptoms/positive experience).

CONTACTS AND LOCATIONS:
Locations (1):
- European Society of Intensive Care medicine, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shanafelt T, Ripp J, Trockel M. Understanding and Addressing Sources of Anxiety Among Health Care Professionals During the COVID-19 Pandemic. JAMA. 2020 Jun 2;323(21):2133-2134. doi: 10.1001/jama.2020.5893. No abstract available. PMID 32259193
- [Result] Shanafelt TD, Boone S, Tan L, Dyrbye LN, Sotile W, Satele D, West CP, Sloan J, Oreskovich MR. Burnout and satisfaction with work-life balance among US physicians relative to the general US population. Arch Intern Med. 2012 Oct 8;172(18):1377-85. doi: 10.1001/archinternmed.2012.3199. PMID 22911330
- [Result] Azoulay E, De Waele J, Ferrer R, Staudinger T, Borkowska M, Povoa P, Iliopoulou K, Artigas A, Schaller SJ, Hari MS, Pellegrini M, Darmon M, Kesecioglu J, Cecconi M; ESICM. Symptoms of burnout in intensive care unit specialists facing the COVID-19 outbreak. Ann Intensive Care. 2020 Aug 8;10(1):110. doi: 10.1186/s13613-020-00722-3. PMID 32770449
- [Result] Azoulay E, Herridge M. Understanding ICU staff burnout: the show must go on. Am J Respir Crit Care Med. 2011 Nov 15;184(10):1099-100. doi: 10.1164/rccm.201109-1638ED. No abstract available. PMID 22086984
- [Result] Aiken LH, Clarke SP, Sloane DM, Sochalski J, Silber JH. Hospital nurse staffing and patient mortality, nurse burnout, and job dissatisfaction. JAMA. 2002 Oct 23-30;288(16):1987-93. doi: 10.1001/jama.288.16.1987. PMID 12387650
- [Result] Dres M, Copin MC, Cariou A, Mathonnet M, Gaillard R, Shanafelt T, Riou B, Darmon M, Azoulay E. Job Strain, Burnout, and Suicidal Ideation in Tenured University Hospital Faculty Staff in France in 2021. JAMA Netw Open. 2023 Mar 1;6(3):e233652. doi: 10.1001/jamanetworkopen.2023.3652. PMID 36976563
- [Result] Azoulay E, Pochard F, Reignier J, Argaud L, Bruneel F, Courbon P, Cariou A, Klouche K, Labbe V, Barbier F, Guitton C, Demoule A, Kouatchet A, Guisset O, Jourdain M, Papazian L, Van Der Meersch G, Reuter D, Souppart V, Resche-Rigon M, Darmon M, Kentish-Barnes N; FAMIREA Study Group. Symptoms of Mental Health Disorders in Critical Care Physicians Facing the Second COVID-19 Wave: A Cross-Sectional Study. Chest. 2021 Sep;160(3):944-955. doi: 10.1016/j.chest.2021.05.023. Epub 2021 May 21. PMID 34023323
- [Result] Azoulay E, Pochard F, Argaud L, Cariou A, Clere-Jehl R, Guisset O, Labbe V, Tamion F, Bruneel F, Jourdain M, Reuter D, Klouche K, Kouatchet A, Souppart V, Lautrette A, Bohe J, Vieillard Baron A, Dellamonica J, Papazian L, Reignier J, Barbier F, Dumas G, Kentish-Barnes N. Resilience and Mental-Health Symptoms in ICU Healthcare Professionals Facing Repeated COVID-19 Waves. Am J Respir Crit Care Med. 2024 Mar 1;209(5):573-583. doi: 10.1164/rccm.202305-0806OC. PMID 38163380
- [Result] Dzau VJ, Kirch DG, Nasca TJ. To Care Is Human - Collectively Confronting the Clinician-Burnout Crisis. N Engl J Med. 2018 Jan 25;378(4):312-314. doi: 10.1056/NEJMp1715127. No abstract available. PMID 29365296
- [Result] West CP, Dyrbye LN, Erwin PJ, Shanafelt TD. Interventions to prevent and reduce physician burnout: a systematic review and meta-analysis. Lancet. 2016 Nov 5;388(10057):2272-2281. doi: 10.1016/S0140-6736(16)31279-X. Epub 2016 Sep 28. PMID 27692469
- [Result] Xu HG, Kynoch K, Tuckett A, Eley R. Effectiveness of interventions to reduce emergency department staff occupational stress and/or burnout: a systematic review. JBI Evid Synth. 2020 Jun;18(6):1156-1188. doi: 10.11124/JBISRIR-D-19-00252. PMID 32813371
- [Result] Quenot JP, Rigaud JP, Prin S, Barbar S, Pavon A, Hamet M, Jacquiot N, Blettery B, Herve C, Charles PE, Moutel G. Suffering among carers working in critical care can be reduced by an intensive communication strategy on end-of-life practices. Intensive Care Med. 2012 Jan;38(1):55-61. doi: 10.1007/s00134-011-2413-z. Epub 2011 Nov 30. PMID 22127481
- [Result] Bienvenu OJ. Is this critical care clinician burned out? Intensive Care Med. 2016 Nov;42(11):1794-1796. doi: 10.1007/s00134-016-4497-y. Epub 2016 Aug 16. No abstract available. PMID 27530295
- [Result] Andersen S, Mintz-Binder R, Sweatt L, Song H. Building nurse resilience in the workplace. Appl Nurs Res. 2021 Jun;59:151433. doi: 10.1016/j.apnr.2021.151433. Epub 2021 Apr 14. PMID 33947518
- [Result] Atay N, Sahin-Bayindir G, Buzlu S, Koc K, Kuyuldar Y. The relationship between posttraumatic growth and psychological resilience of nurses working at the pandemic clinics. Int J Nurs Knowl. 2023 Jul;34(3):226-235. doi: 10.1111/2047-3095.12397. Epub 2022 Oct 27. PMID 36303467
- [Result] Sadeghi Avval Shahr H, Yazdani S, Afshar L. Professional socialization: an analytical definition. J Med Ethics Hist Med. 2019 Dec 7;12:17. doi: 10.18502/jmehm.v12i17.2016. eCollection 2019. PMID 32328230
- [Result] McAleer P, Todorov A, Belin P. How do you say 'hello'? Personality impressions from brief novel voices. PLoS One. 2014 Mar 12;9(3):e90779. doi: 10.1371/journal.pone.0090779. eCollection 2014. PMID 24622283
- [Derived] Azoulay E, Myatra SN, Heras La Calle G, Jaber S, Boulanger C, Demirkyran O, Theodorakopoulou M, Paiva JA, Arabi YM, Burghi G, van Heerden PV, Al Fares A, Kentish-Barnes N, Martin-Delgado MC, Mistraletti G, Francois G, Barth A, De Waele J, Shanafelt TD, Darmon M, Cecconi M; European Society of Intensive Care Medicine. Positive communication for decreasing burnout in intensive-care-unit staff: a cluster-randomized trial. Intensive Care Med. 2025 Nov;51(11):2031-2041. doi: 10.1007/s00134-025-08134-2. Epub 2025 Oct 30. PMID 41165789
- [Derived] Azoulay E, Barnes NK, Myatra SN, Delgado MM, Arabi Y, Boulanger C, Mistraletti G, Theodorakopoulou M, Van Heerden V, Paiva JA, Demirkyran O, La Calle GH, Al Fares A, Burghi G, Francois G, Barth A, De Waele J, Jaber S, Darmon M, Cecconi M. HELLO: a protocol for a cluster randomized controlled trial to enhance interpersonal relationships and team cohesion among ICU healthcare professionals. Intensive Care Med Exp. 2024 Oct 7;12(1):90. doi: 10.1186/s40635-024-00677-w. PMID 39373831